CLINICAL TRIAL: NCT02583737
Title: Histological and Microtomographic Comparative Study Between Lyophilized or Frozen Bone Allografts for Sinus-lifting: A Randomized Clinical Trial
Brief Title: Comparative Study Between Lyophilized or Frozen Bone Allografts for Sinus-lifting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria Cristina Zindel Deboni, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAEE 30738714.0.0000.0075.
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Disorder of Maxillary Sinus; Accessory; Bone; Bone Atrophy
Keywords: bone; maxillary sinus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group lyophilized bone allograft (Active Comparator): sinus lifting with tissue bank lyophilized bone filling
  Interventions: Procedure: lyophilized bone allograft
- group freeze bone allograft (Active Comparator): sinus lifting with freeze bone bank filling
  Interventions: Procedure: freeze bone allograft

INTERVENTIONS:
Procedure: freeze bone allograft — sinus lifting filling procedure employing freeze bone allograft from tissue bone bank.
  Arms: group freeze bone allograft
Procedure: lyophilized bone allograft — sinus lifting filling procedure employing lyophilized bone allograft from tissue bone bank.
  Arms: group lyophilized bone allograft

SUMMARY:
Bone resorption and atrophy in maxillary posterior region is due to severe periodontal disease and is consequent tooth extractions. Sinus pneumatisation can occur after tooth extraction and alveolar bone loss. Consequently, bone-reducing volume at that region is a great challenge to implantodontists. Sinus lifting surgery have been practiced since 80's and many biomaterials have been used to solve filling issues to maintain the sinus floor lifted in a position that can allow dental implants installation. Bone grafts have shown to be the best choice of filling grafts. Despite autologous bone are the gold standard filling biomaterial it is associates with great mortality and morbidity. So, bone allografts from tissue bank had been shown to be an advantageous alternative. Lyophilized or freeze tissue bone are the most common allografts but literature is poor in randomized controlled parallel clinical trials regarding those filling grafts for sinus lifting. The aim of this study is to perform a randomized controlled clinical trial comparing two bone allografts: lyophilized and freeze bone allografts from human bone tissue bank. The investigators want to verify which one can develop greater osteogenesis, if is there any difference between them regarding the architectural trabeculae formation, if there are different patterns of reabsorption and finally if is there any differences between them regarding primary and lately dental implants stability. To answer those questions the investigators propose firstly, to carry out microtomographic and histological analysis from trephine bone samples after six months of sinus lifting and grafting in healthy participants undergoing osseointegrated dental implants. Secondly, the primary and lately implant stability is going to be achieved employing Resonance Frequency Analysis (RFA).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* totally or partially edentulous patients, bilaterally, in upper premolar or molar region; presenting maxillary sinus lifting necessity with bilateral alveolar bone height lower than 5mm and indication for at least one osseointegrated dental implant in premolar or molar region.

Exclusion Criteria:

* recent sinusitis history
* hypersensibility for sinus allergens, tabagism, ethylism
* severe periodontal disease, diabetes, hypertension.
* Cases that occur schneiderian membrane perforation will be excluded from the final sample.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
volume of bone neoformation in mm3 | six months after grafting
  computational software for analysis the micro CT scanning of trephine bone samples images
area of bone neoformation in μm2 | six months after grafting
  IMAGEJ histomorphometric software for analysis of trephine bone samples micrographic images

SECONDARY OUTCOMES:
dental implants stability value | six months after grafting
  primary implant stability by Resonance Frequency Analysis (RFA) in ISQ
dental implants stability value | six months after dental implant
  late stability by Resonance Frequency analysis (RFA) in ISQ

REFERENCES:
- [Background] Acocella A, Bertolai R, Nissan J, Sacco R. Clinical, histological and histomorphometrical study of maxillary sinus augmentation using cortico-cancellous fresh frozen bone chips. J Craniomaxillofac Surg. 2011 Apr;39(3):192-9. doi: 10.1016/j.jcms.2010.03.019. Epub 2010 May 7. PMID 20452232
- [Background] Chiapasco M, Giammattei M, Carmagnola D, Autelitano L, Rabbiosi D, Dellavia C. Iliac crest fresh-frozen allografts and autografts in maxillary and mandibular reconstruction: a histologic and histomorphometric evaluation. Minerva Stomatol. 2013 Jan-Feb;62(1-2):3-16. English, Italian. PMID 23422679
- [Background] de Castilho TR, Tortamano P, Marotti J, de Andrade JC Jr, Chilvarquer I, Ximenez ME, Alves MT. Clinical and Histomorphometric Evaluation of Fresh Frozen Bone Allograft in Sinus Lift Surgery. Clin Implant Dent Relat Res. 2016 Feb;18(1):40-50. doi: 10.1111/cid.12234. Epub 2014 Jun 6. PMID 24909241
- [Background] Deluiz D, Oliveira LS, Pires FR, Tinoco EM. Time-dependent changes in fresh-frozen bone block grafts: tomographic, histologic, and histomorphometric findings. Clin Implant Dent Relat Res. 2015 Apr;17(2):296-306. doi: 10.1111/cid.12108. Epub 2013 Jul 9. PMID 23837530
- [Background] Eskan MA, Greenwell H, Hill M, Morton D, Vidal R, Shumway B, Girouard ME. Platelet-rich plasma-assisted guided bone regeneration for ridge augmentation: a randomized, controlled clinical trial. J Periodontol. 2014 May;85(5):661-8. doi: 10.1902/jop.2013.130260. Epub 2013 Jul 29. PMID 23895252
- [Background] Goulet JA, Senunas LE, DeSilva GL, Greenfield ML. Autogenous iliac crest bone graft. Complications and functional assessment. Clin Orthop Relat Res. 1997 Jun;(339):76-81. doi: 10.1097/00003086-199706000-00011. PMID 9186204
- [Background] Holtzclaw D, Toscano N, Eisenlohr L, Callan D. The safety of bone allografts used in dentistry: a review. J Am Dent Assoc. 2008 Sep;139(9):1192-9. doi: 10.14219/jada.archive.2008.0334. PMID 18762629
- [Background] Le B, Rohrer MD, Prasad HS. Screw "tent-pole" grafting technique for reconstruction of large vertical alveolar ridge defects using human mineralized allograft for implant site preparation. J Oral Maxillofac Surg. 2010 Feb;68(2):428-35. doi: 10.1016/j.joms.2009.04.059. Epub 2010 Jan 15. PMID 20116718
- [Background] Pimentel AC, Napimoga MH, Manzi MR, Sendyk WR. Reconstruction of the edentulous mandible with fresh frozen bone grafts and implants: a 4-year report of a prospective clinical study. Cell Tissue Bank. 2014 Mar;15(1):1-6. doi: 10.1007/s10561-012-9352-y. Epub 2012 Nov 27. PMID 23184222
- [Background] Pelegrine AA, Sorgi da Costa CE, Sendyk WR, Gromatzky A. The comparative analysis of homologous fresh frozen bone and autogenous bone graft, associated or not with autogenous bone marrow, in rabbit calvaria: a clinical and histomorphometric study. Cell Tissue Bank. 2011 Aug;12(3):171-84. doi: 10.1007/s10561-010-9178-4. Epub 2010 May 16. PMID 20473718
- [Background] Schwartz Z, Goldstein M, Raviv E, Hirsch A, Ranly DM, Boyan BD. Clinical evaluation of demineralized bone allograft in a hyaluronic acid carrier for sinus lift augmentation in humans: a computed tomography and histomorphometric study. Clin Oral Implants Res. 2007 Apr;18(2):204-11. doi: 10.1111/j.1600-0501.2006.01303.x. PMID 17348885